CLINICAL TRIAL: NCT01681589
Title: Relationship Between Attention and Emotional Regulation Post-TBI: Probing Neural Circuitry With Transcranial Direct Current Stimulation
Brief Title: Relationship Between Attention and Emotional Regulation Post-Traumatic Brain Injury (TBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-00685
Record Dates: First submitted 2012-08-16; First posted 2012-09-10 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Traumatic Brain Injury; Rehabilitation; Therapy
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Control Group (Sham Comparator): The control group will receive sham-tDCS and computerized cognitive training also twice a week for 20 minutes for 6 weeks (12 training sessions).
  Interventions: Device: Control Group
- Transcranial Direct Current Stimulator (TDCS) (Experimental): The experimental group will receive active tDCS for 20 minutes and computerized cognitive training twice a week for 30 minutes for 6 weeks.
  Interventions: Device: Transcranial Direct Current Stimulator (TDCS)
- Healthy Control Group (Other): Fifteen (15) healthy control subjects will participate.
  Interventions: Other: Healthy Control Group

INTERVENTIONS:
Device: Transcranial Direct Current Stimulator (TDCS) — Group will receive active TDCS
  Other Names: Fisher Wallace Cranial Stimulator; The Fisher Wallace Stimulator, Model FW-100; FDA 510 (K)Cleared number K903654
  Arms: Transcranial Direct Current Stimulator (TDCS)
Device: Control Group — This group will receive Sham TDCS
  Arms: Control Group
Other: Healthy Control Group — Healthy Controls will be involved in the Study. Healthy Controls will receive no Intervention. There will be 1 screening visit and 1 testing visits.
  Arms: Healthy Control Group

SUMMARY:
The purpose of this pilot study is to investigate the relationship between attention and emotional function post-Traumatic Brain Injury (TBI) in an effort to better understand the cognitive mechanisms of emotional processing in patients with TBI, and explore novel treatment strategies to improve emotional regulation using with transcranial direct current stimulation (tDCS) to modulate activity in the dysfunctional prefrontal-limbic circuits.

DETAILED DESCRIPTION:
Thirty (30) individuals status post TBI with complaints of emotional dysfunction 6 months post-brain injury and Fifteen (15) healthy controls will participate in the study. The experimental group will receive active tDCS for 20 minutes and computerized cognitive training twice a week for 30-45 minutes for 6 weeks as described below. The control group will receive sham-tDCS 20 minutes and computerized cognitive training for 30-45 minutes twice a week for 6 weeks (12 training sessions). The sham group will not receive real tDCS after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Brain Injury at least 6 months prior
* Family or self-identification of cognitive or emotional difficulties
* Unchanged and stabilized medical treatment in the three weeks prior to the screening

Exclusion Criteria:

* Any social or medical problem that precludes completion of the protocol.
* Presence of focal motor deficits in the upper extremities.
* Comorbid psychiatric disease such as schizophrenia, or active substance abusers (except nicotine).
* History of craniectomy, active infection, or seizure activity beyond 1 week post-TBI.
* Complicating medical problems such as uncontrolled hypertension, diabetes with signs of neuropathy, and previous neurological illness such as head trauma, prior stroke, epilepsy or demyelinating disease, implanted neuromodulatory or electronic device, metal in head
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prin Amorapanth, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. Data transfer was not ideal, and no study data are available.
Period: Overall Study
Arm/Group | Control Group | Transcranial Direct Current Stimulator (TDCS) | Healthy Control Group
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. Data transfer was not ideal, and no study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Transcranial Direct Current Stimulator (TDCS) | Healthy Control Group | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Baseline Measures Before Treatment
Description: Patients meeting criteria to particpate in the study will be tested at baseline. During Visit 1, patients will be tested to measure how alert they are, their ability to perform actions one after the other and other mental functions. On Visit 2, patients will be tested on your ability to control your emotions. On Visit 3, patients will have a brain scan (MRI) to help the investigators understand how various parts of your brain are connected.
Time Frame: Week 1
Population: as for baseline characteristics
Arm/Group | Control Group | Transcranial Direct Current Stimulator (TDCS) | Healthy Control Group
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Post Treatment Measures to Check Improvements
Description: Testing will be done again at the end of 6 weeks. This will allow the investigators to determine if there have been improvements in the patients attention and emotional function. The same assessments will be repeated again as with Visits 1-3. Investigators will ask questions regarding patients emotional well-being. An MRI will once again be performed.
Time Frame: Week 8
Population: as for baseline characteristics
Arm/Group | Control Group | Transcranial Direct Current Stimulator (TDCS) | Healthy Control Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 years
Description: The PI and study team has left the institution. Efforts were made to contact the PI/study team members, but were unsuccessful. Data transfer was not ideal, and no study data are available.
Arm/Group | Control Group | Transcranial Direct Current Stimulator (TDCS) | Healthy Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT01681589/Prot_000.pdf